CLINICAL TRIAL: NCT01495182
Title: A Double-blind, Randomized, Crossover Trial to Assess the Gastrointestinal Tolerability of a Dietary Fiber Ingredient in Healthy Men and Women
Brief Title: Effects of Dietary Fiber on Gastrointestinal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2011-12-14; First posted 2011-12-19 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2011-12

CONDITIONS: Gastrointestinal Health
Keywords: Dietary fiber; Gastrointestinal toleration; Fecal weight
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dietary Fiber - Dose 1 (Experimental): Dietary fiber will be added to study foods
  Interventions: Other: Dietary fiber
- Dietary Fiber - Dose 2 (Experimental): Dietary fiber will be added to study foods
  Interventions: Other: Dietary fiber
- Control (Active Comparator): Study foods with no added fiber will be given
  Interventions: Other: Dietary fiber

INTERVENTIONS:
Other: Dietary fiber — A proprietary fiber will be given to subjects

SUMMARY:
The purpose of the study will be to assess the gastrointestinal effects of a dietary fiber in healthy, adult volunteers.

DETAILED DESCRIPTION:
The study is a blinded, cross-over design with subjects completing three, two-week treatment periods, separated by two, two-week washouts. Volunteers will consume a dietary fiber for two of the treatment periods at two dose levels. The fiber will be added to foods and dispensed to subjects to be consumed twice a day during each treatment period. During the control period, subjects will receive the same study foods, but with no added fiber. Major outcomes will include fecal weight, and responses to questionnaires that assess fecal characteristics, bowel habits and gastrointestinal tolerability.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* age 18 - 54 years
* BMI < 30 kg/m2

Exclusion Criteria:

* presence of GI or other serious diseases known to affect GI function
* recent use of antibiotics
* very high fiber intake
* use of medications known to affect GI function
* presence of allergies to study foods

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerability | subjects will report weekly for 6 weeks
  Questionnaire to assess symptoms such as nausea, bloating, and flatulence

SECONDARY OUTCOMES:
Fecal output | subjects will collect fecal output for 12 days within a six-week period
  Fecal weight and stool characteristics will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Principal Investigator — Provident Clinical Research Center
Locations (1):
- Provident Clinical Research and Consulting Inc, Glen Ellyn, Illinois, United States